CLINICAL TRIAL: NCT05405530
Title: Nasal Mask Oxygen Reduces the Incidence of Hypoxia Undergoing Gastrointestinal Endoscopy Under Propofol Sedation: a Multicenter Randomized Controlled Trial
Brief Title: Nasal Mask Kit in Gastrointestinal Endoscopy
Acronym: NASO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Henan Provincial People's Hospital (Other); First Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, diansan su, Vice Chair of the Department of Anesthesiology, RenJi Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RenJiH-2022-01-04
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Hypoxia; Gastric Cancer; Gastric Polyp; Colon Polyp; Colon Cancer; Esophageal Cancer
Keywords: nasal mask; Hypoxia; Gastrointestinal endoscopy; Propofol; Capnographic Monitoring
MeSH Terms: conditions — Hypoxia; Stomach Neoplasms; Polyposis, Gastric; Colonic Polyps; Colonic Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- nasal mask oxygen group (Experimental): In this group, patients use the nasal mask oxygen kit for oxygenation.
  Interventions: Device: nasal mask oxygen kit
- regular nasal cannula group (Active Comparator): In this group, patients use the regular nasal cannula for oxygenation.
  Interventions: Device: regular nasal cannula

INTERVENTIONS:
Device: nasal mask oxygen kit — Using the nasal mask oxygen kit for oxygenation.
  Arms: nasal mask oxygen group
Device: regular nasal cannula — Using nasal cannula for oxygenation.
  Arms: regular nasal cannula group

SUMMARY:
Hypoxia is the most common adverse event in gastrointestinal endoscopes sedated with propofol. The nasal mask oxygen kit has good sealing to ensure an adequate oxygen supply and is convenient and economical.The aim of this randomized study was to determine whether the nasal mask oxygen kit reduces the incidence of hypoxia in gastrointestinal endoscopes procedures.

ELIGIBILITY:
Inclusion Criteria:

* 18≤ Age ≤60
* patients undergoing combined gastroendoscopy and colonoscopy procedure
* patients signed informed consent form
* ASA classification I-II
* Estimated procedure time <=45min

Exclusion Criteria:

* Coagulation disorders or a tendency of nose bleeding
* Diagnosed heart disease (heart failure, angina, myocardial infarction, arrhythmia, etc.)
* Diagnosed chronic obstructive pulmonary disease or current other acute or chronic lung disease requiring supplemental chronic or intermittent oxygen therapy)
* hypoxia (SpO2< 90 % )
* Upper respiratory tract infection
* increased intracranial pressure
* Fever (core body temperature >37.5 ℃)
* Pregnancy, breastfeeding, or positive pregnancy test
* Emergency procedure or surgery
* Multiple trauma
* Allergy to propofol or tape and adhesives
* BMI<18.5 or BMI>30

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1204 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
The incidence of hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours]
  (75% ≤ SpO2 < 90% for <60 s)

SECONDARY OUTCOMES:
The incidence of sub-clinical respiratory depression | Patients will be followed for the duration of hospital stay, an expected average about 2 hours]
  (90% ≤ SpO2 < 95%)
The incidence of severe hypoxia | Patients will be followed for the duration of hospital stay, an expected average about 2 hours
  (SpO2 < 75% or 75% ≤ SpO2 < 90% for >/=60 s)
The incidence of other adverse events | Patients will be followed for the duration of hospital stay, an expected average about 2 hours]
  Other adverse events recorded by tools proposed by the World Society of Intravenous Anesthesia International Sedation Task Force

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Renji Hospital, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3months and ending 5 years following article publication.
Access Criteria: The data will be available to other researchers upon request, with information shared after approval by the corresponding author (D-SS).

REFERENCES:
- [Derived] Cheng X, Zhang X, Zhang J, Hu Z, Zhang J, Lian Q, Ding X, He Y, Shi M, Zhang Y, Tian M, Zheng H, Li Z, Wang Y, Yu W, Shao J, Su D. Efficacy of a nasal mask oxygen kit versus regular nasal cannula in sedated gastrointestinal endoscopy: a multicentre, randomised clinical trial. BMJ Open Gastroenterol. 2025 Jul 7;12(1):e001834. doi: 10.1136/bmjgast-2025-001834. PMID 40623715